CLINICAL TRIAL: NCT06876831
Title: Inpatient Capture: A Mixed Methods Study to Develop an Inpatient Lung Cancer Screening Program in a Safety Net Hospital.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Physician Affiliate Group of New York (Other)
Collaborators: Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Natoushka Trenard, Attending physician, MD MPH, Physician Affiliate Group of New York
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 23-02-006-182
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer Screening Program

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meets LCS criteria and former smoker (Experimental): LDCT on discharge, scheduled date of LDCT, or Lung cancer screening referral
  Interventions: Other: Shared decision making for LDCT (3 potential outcomes LDCT on discharge, scheduled date of LDCT, or Lung Cancer Screening referral)
- Meets LCS criteria and active smoker (Experimental): Inpatient LCS SDM (potential outcomes: 1- LDCT on discharge, 2-scheduled date of LDCT, 3-LCS referral. Along with Inpatient Tobacco Cessation/Reduction Counseling (Handouts, NYC Quits number, medication recommendations to primary team).
  Interventions: Other: Shared decision making for LDCT (3 potential outcomes LDCT on discharge, scheduled date of LDCT, or Lung Cancer Screening referral); Behavioral: Inpatient Tobacco Cessation Counseling (Handouts, NYC Quits number, Medication Recommendations to primary team, Smoking cessation referral)

INTERVENTIONS:
Other: Shared decision making for LDCT (3 potential outcomes LDCT on discharge, scheduled date of LDCT, or Lung Cancer Screening referral) — These interventions will be facilitated as an inpatient
Behavioral: Inpatient Tobacco Cessation Counseling (Handouts, NYC Quits number, Medication Recommendations to primary team, Smoking cessation referral) — Active smokers only will received inpatient tobacco cessation counseling/risk reduction
  Arms: Meets LCS criteria and active smoker

SUMMARY:
Lung cancer continues to be the leading cause of cancer death in the United States. There are several important disparities in lung cancer mortality: racial and ethnic minorities, those with serious mental illness and those with lower socioeconomic status experience higher lung cancer mortality compared to the general population. Lung cancer screening (LCS) with annual low dose chest CT can reduce lung cancer mortality by 20% for high-risk patients, but has been generally underutilized with uptake of 5-15% by eligible patients across the United States. Half of all patients eligible for LCS remain current smokers, and the additional benefits of tobacco cessation services can increase the benefits of LCS clinical encounters in these patients. Despite the proven benefit of LCS and tobacco cessation, it remains out of reach for many with barriers across the patient, provider, and health-care system levels with resultant disparities in uptake of LCS and effective tobacco cessation that may exaggerate disparities in clinical lung cancer early detection and mortality. The majority of LCS care occurs across several visits in an outpatient clinical setting, which may make it inaccessible to the most vulnerable patients.

Our central objective is to extend the reach of lung cancer and tobacco screening through the implementation and evaluation of a program extending these services inpatient in a public hospital that serves a known high-risk and diverse population in East Harlem. Preliminary data obtained from a retrospective quality improvement project examined data from patients admitted over a 3 month period in early 2022. Of 1374 unique patients were admitted to our hospital, 112 patients met LCS eligibility criteria and over 80% had no evidence of having been screened. Forty-seven percent identified as Black and 33.9% as Hispanic, groups known to have worse lung cancer outcomes. While smoking data was incomplete on a majority of patients, 75% of all inpatient admissions were noted to be currently smoking. This, our preliminary data suggest that an inpatient program to provide smoking cessation and LCS in a safety-net hospital may be an effective tool to increase the reach of LCS in a known high-risk demographic and address disparities in LCS and tobacco cessation services.

This proposal represents a prospective pilot study to develop, implement and evaluate an inpatient LCS and tobacco cessation program.

ELIGIBILITY:
Inclusion Criteria:

* 50-80 years of age
* greater than or equal to 20 pack year history
* currently smoking or have quit within the last 15 years

Exclusion Criteria:

* < 50 years of age, > 80 years of age
* < 20 pack year history
* quit smoking greater than 15 years

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
up-to-date status on LCS at 3 months of hospital discharge | 3 months post hospital discharge
  Up-to-date status is defined as the completion of a low-dose chest CT within 15 months. Estimating equations will also be used to determine the independent association of the intervention with increase in prevalence of up-to-date LCS adjusted for patient demographic features and underlying time-trends.

SECONDARY OUTCOMES:
difference in referrals for LCS and completion of smoking cessation/LCS eligibility data | 6 months
  Differences in proportions will be used to compare the prevalence of up-to-date LCS between pre and post period.

CONTACTS AND LOCATIONS:
Locations (1):
- Metropolitan Hospital/ NYCHHC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be collected and de-identified for analysis. Only analysis of de-identified data will be shared.